CLINICAL TRIAL: NCT03148548
Title: Iliofemoral Thrombosis and Postthrombotic Syndrome: Registration and Analysis Within the Frankfurt Thrombophilia Registry
Brief Title: Substudy - Evaluation of Patients With Iliac Vein Thrombosis
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Sponsor
Other Study IDs: ILIACA-PTS
Record Dates: First submitted 2017-03-07; First posted 2017-05-11 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Iliac Vein Thrombosis
Keywords: VTE; thrombophilia screening; patients; risk factors; post-thrombotic syndrome
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — whole blodd, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with iliofermoral thrombosis without rekanalisation: subjects with proven iliofemoral thrombosis (V. cava-aplasia, pelvic vein thrombosis, VTE) which was proven by objective methods such as Duplex sonography, CT/MRT, phlebography and who did not undergo recanalisation
  Interventions: Genetic: thrombophilia screening
- Patients with ilifermoral thrombosis with rekanalisation: subjects with proven iliofemoral thrombosis (V. cava-aplasia, pelvic vein thrombosis, VTE) which was proven by objective methods such as Duplex sonography, CT/MRT, phlebography and who did undergo recanalisation
  Interventions: Genetic: thrombophilia screening

INTERVENTIONS:
Genetic: thrombophilia screening — genetic Evaluation of Factor-V-Leiden, Factor-II_G20210A Mutation;

SUMMARY:
Patients with previous diagnosis of iliac vein thrombosis are enrolled in this registry. Using standardized questionnaire, clinical data detailing venous thromboembolism and contributing VTE risk factors are recorded. Results of technical and laboratory investigations including screening of thrombophilic disorders were additionally entered into the database.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* subjects with iliofermoral thrombosis, which has been proven by objective measurements (Duplex sonography, phlebography, CT/MRT) later than 1996

Exclusion Criteria:

* <18 years
* > 80 years
* surface or deep vein thrombosis without affection of pelvis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with previous iliofermoral thrombosis, which has been proven by objective measurements (Duplex sonography, phlebography, CT/MRT)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of postthrombotic Syndrome after iliofemoral thrombosis | up to 20 years after occurrence of iliofemoral thrombosis
  The incidence and severity of postthrombotic Syndrome will be measured by te VILALLTA-Score

SECONDARY OUTCOMES:
Distribution of gender in Iliofemoral thrombosis | since 1996
  Distribution of gender (man or woman)
Distribution of affected side in Iliofemoral thrombosis | since 1996
  distribution of affected side (left or right side)
Disease-specific quality of life instrument for use in venous diseases of the leg (VEINES-QOL) | 1 year
  A quality of life questionaire comprises 25 items that quantify disease effect on quality of life
Incidence of venous claudication | 1 year
  Walking distance on treadmill

CONTACTS AND LOCATIONS:
Overall Officials: Edelgard Lindhoff-Last, Prof., Principal Investigator — Cardioangiologisches Centrum Bethanien
Locations (1):
- Cardioangiologisches Centrum Bethanien, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No